CLINICAL TRIAL: NCT07117435
Title: A Phase Ib/III Study to Evaluate the Safety and Efficacy of Paclitaxel Cationic Liposome (Hepatic Arterial Infusion) in Combination With Systemic Therapy as First-Line Treatment in Colorectal Liver Metastases
Brief Title: Paclitaxel Cationic Liposome (Hepatic Arterial Infusion) in Combination With Systemic Therapy as First-Line Treatment in Colorectal Liver Metastases
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HA131-004
Record Dates: First submitted 2025-08-05; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Colorectal Liver Metastases; First-line Treatment
MeSH Terms: interventions — Injections; Oxaliplatin; Capecitabine; Bevacizumab

STUDY DESIGN:
Intervention Model Description: All participants receive the same treatment, and there is no comparison group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental arm (Experimental): Paclitaxel cationic liposome was administered via hepatic arterial infusion on Day 15 of each 3-week cycle, and in a gradual increment dose range from 33 mg/m^2 to 55 mg/m^2, combined with systemic therapy (Oxaliplatin, Capecitabine, with or without Bevacizumab)
  Interventions: Drug: paclitaxel cationic liposome for injection; Drug: Oxaliplatin; Drug: Capecitabine; Drug: Bevacizumab

INTERVENTIONS:
Drug: paclitaxel cationic liposome for injection — Paclitaxel cationic liposome was administered through hepatic arterial catheter infusion, in a gradual increment dose range from 33 mg/m^2 to 55 mg/m^2
Drug: Oxaliplatin — Oxaliplatin 130 mg/m2 i.v. on D1
Drug: Capecitabine — Capecitabine 1000 mg/m2 p.o. Bid on Day 1-14
Drug: Bevacizumab — Bevacizumab 7.5 mg/kg i.v. on D1

SUMMARY:
This is a phase Ib/III, randomized, multicenter study evaluating the efficacy and safety of hepatic arterial infusion of paclitaxel cationic liposome in combination with systemic therapy (Oxaliplatin, Capecitabine, with or without Bevacizumab) as first-line treatment in colorectal liver metastases.

DETAILED DESCRIPTION:
This study includes 2 parts. In Phase Ib part of this study, paclitaxel cationic liposome was administered via hepatic arterial infusion on Day 15 of each 3-week cycle, and in a gradual increment dose from the low-level to the high-level, with the first cycle (21 days) being the DLT observation period. In the Phase III part of this study, participants will be randomized in 1:1 ratio to receive either hepatic arterial infusion of paclitaxel cationic liposome (at the dose to be determined in the Phase Ib) in combination with systemic therapy or systemic therapy.

The primary purpose of the Phase Ib part of this study is to determine the recommended Phase III dose (RP3D) of paclitaxel cationic liposome administered via hepatic arterial infusion on Day 15 of each 3-week cycle.

The primary purpose of the Phase III part of this study is to measure the efficacy and safety of hepatic arterial infusion of paclitaxel cationic liposome in combination with systemic therapy (Oxaliplatin, Capecitabine, with or without Bevacizumab) as first-line treatment in colorectal liver metastases.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age range: 18 - 75 years old (inclusive), gender not limited.
* 2. For patients with colorectal liver metastases have been histologically or cytologically confirmed and who are assessed by multidisciplinary team (MDT) to be inoperable for radical surgical resection:

  1. Have not received systemic treatment for the metastatic or recurrent disease;
  2. For patients who have received neoadjuvant/adjuvant therapy before, the time interval between the last administration and disease progression must be ≥ 6 months;
  3. Allow patients who have received local treatment and progressed.
* 3. According to RECIST v1.1, at least one measurable lesion in the hepatic arterial infusion area (long diameter ≥ 1 cm and no previous local treatment).
* 4. Eastern Cooperative Oncology Group (ECOG) performance status score of 0-1.
* 5. Life expectancy of at least 3 months.
* 6. Adequate organ function, with laboratory tests meeting the following criteria (no blood transfusion or hematopoietic growth factors within 14 days)
* 7. Fertile patients (male and female) must agree to use reliable contraceptive methods (hormonal contraceptives, barrier methods, or abstinence) with their partners during the study and for at least 6 months after the last dose of study intervention. Women of childbearing potential must have a negative pregnancy test within 7 days prior to enrollment.
* 8. Fully understand the clinical study and voluntarily sign a written informed consent form.

Exclusion Criteria:

* 1. Patients known to have microsatellite instability high (MSI-H) or mismatch repair deficiency (dMMR), and have been evaluated by the investigators to be eligible for immune checkpoint inhibitor therapy.
* 2. Patients known to have wild-type RAS and BRAF, and have been evaluated by the investigators to be eligible for anti-epidermal growth factor receptor (EGFR) drug therapy.
* 3. Unresolved adverse reactions from previous anti-tumor treatments not yet recovered to CTCAE 5.0 grade ≤ 1 (except for alopecia or other toxicities deemed non-risky by the investigators).
* 4. Central nervous system metastasis with clinical symptoms, or meningeal metastasis, or there are other evidences indicating that the patient's central nervous system metastasis or meningeal metastatic lesions have not been controlled, and the investigators judges that the patient is not suitable for enrollment.
* 5. Patients with contraindications for transcatheter arterial infusion.
* 6. Patients with active infections within 2 weeks prior to administration (NCI CTC AE v5.0 ≥ grade 2) (Defined as requiring intravenous administration of antibacterial, antifungal or antiviral drugs for treatment).
* 7. Patients with grade 2 or above peripheral neuropathy (NCI CTC AE v5.0).
* 8. Patients with a history of autoimmune diseases, immunodeficiency disorders, including HIV positive test results, or suffering from other acquired or congenital immune deficiencies, or those currently using immunosuppressive agents.
* 9. Hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) positive with HBV DNA ≥ 2×103 IU/mL (can use continuous antiviral treatment); or anti-hepatitis C virus antibody (HCV-Ab) positive with HCV RNA above the measurable limit; or active syphilis.
* 10. Patients with known contraindications to capecitabine or oxaliplatin, paclitaxel or cationic liposome, or have severe allergic reactions; note: If the subject has contraindications to bevacizumab or has severe allergic reactions to any component of bevacizumab, it will not affect the enrollment but should not use bevacizumab in the study, and the specific reasons need to be recorded.
* 11. Patients need to receive strong inducers and strong inhibitors of CYP2C8 and CYP3A4 within 2 weeks before the first study treatment or during the treatment.
* 12. Patients had or have non-infectious pneumonia/interstitial lung disease that requires systemic glucocorticoid treatment.
* 13. Severe cardiovascular disease history, including but not limited to:

  * Long QT syndrome;
  * High-degree atrioventricular block;
  * Severe arrhythmia that is not well controlled by medication;
  * Chronic heart failure history and NYHA cardiac function classification ≥ 3;
  * Severe valvular regurgitation or stenosis that requires treatment;
  * Acute coronary syndrome or severe myocardial disease within 6 months before screening;
  * Uncontrolled hypertension;
  * Echocardiography suggests LVEF < 50%;
* 14. Patients with a previous history of severe neurological or mental disorders (including epilepsy or dementia) lead to compliance issues.
* 15. Patients with ultrasound-detected limb vascular thrombosis with potentially serious consequences during screening, or who with thromboembolic events within 3 months prior to enrollment.
* 16. Patients with a history of severe bleeding, or who experienced major bleeding events such as intracranial hemorrhage, gastrointestinal bleeding, or purpura within the last 3 months.
* 17. Any other reasons deemed by the investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Estimated)
Dates: Start 2025-05-13 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
The incidence of dose-limiting toxicity（DLT ） | The first Cycle(21 days)
Incidence and severity of AEs and SAEs (according to NCI-CTCAE 5.0) | Up to approximately 1 years

SECONDARY OUTCOMES:
AUC0-t | The first four cycles ( each cycle is 21 days)
AUC0-∞ | The first four cycles ( each cycle is 21 days)
Cmax | The first four cycles ( each cycle is 21 days)
Kel | The first four cycles ( each cycle is 21 days)
Tmax | The first four cycles ( each cycle is 21 days)
Vz | The first four cycles ( each cycle is 21 days)
t1/2 | The first four cycles ( each cycle is 21 days)
CL | The first four cycles ( each cycle is 21 days)
Overall response rate（ORR） | Up to approximately 1 years
Disease control rate（DCR） | Up to approximately 1 years
Duration of Response（DoR） | Up to approximately 1 years
Progression-Free-Survival（PFS） | Up to approximately 2 years
Time to Progression（TTP） | Up to approximately 2 years
Overall survival（OS） | Up to approximately 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Sun Yat-sen University，Lishui Central Hospital, Lishui, Zhejiang, China